CLINICAL TRIAL: NCT02291588
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AMG 811 in Subjects With Systemic Lupus Erythematosus
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AMG 811 in Subjects With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20060203
Record Dates: First submitted 2014-11-03; First posted 2014-11-14 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — AMG 811

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMG 811 (Experimental): AMG 811 administered as subcutaneous and intravenous doses
  Interventions: Drug: AMG 811
- Placebo (Placebo Comparator): No active drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 811 — A single dose of AMG 811 or placebo will be adminstered.
  Arms: AMG 811
Drug: Placebo — contains no active drug
  Arms: Placebo

SUMMARY:
This first-in-human, multicenter study to evaluate the administration of placebo or AMG 811 single subcutaneous and intravenous dose to subjects with SLE

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE ncluding a positive antinuclear antibodies (ANA) test at least 6 months before randomization; any concurrent SLE pharmacologic regimen (including leflunomide, methotrexate, and anti-malarials) was stable for at least 30 days before randomization; prednisone ≤ 20 mg/day (or equivalent) was permitted; 1 increase or decrease of ≤ 5mg/day prednisone equivalent was allowed within 30 days before randomization

Exclusion Criteria:

* Subjects who, in the clinical judgment of the investigator, had severe disease; subject who had at least 1 BILAG 'A' score or 2 BILAG 'B' scores in any of the organ systems at screening; signs or symptoms of a viral or bacterial infection within 30 days of study randomization, or recent history of repeated infections, evidence of liver disease; concurrent receipt of mycophenolate mofetil or azathioprine; prior administration of another biologic that primarily targets the immune system within 1 year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-12; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as measured by subject incident of treatment-emergent adverse events, clinically significant changes in vital signs, physical examination endpoints, clinical laboratory safety tests, and ECGs | between 84 and 196 days
  Subject incidence of treatment-emergent adverse events, clinically significant changes in vital signs, physical examination endpoints, clinical laboratory safety tests, and ECGs

SECONDARY OUTCOMES:
Pharmacokinetic profile of AMG 811 including tmax, AUClast and Cmax | between 84 and 196 days
  Serum concentration and derived PK parameters

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com